CLINICAL TRIAL: NCT00005524
Title: Mental Stress, Autonomic Function, and Heart Disease
Status: Completed | Type: Observational
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5051; R01HL059332 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2005-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To examine the vagal, vascular sympathetic, and mechno-structural components of baroreflex regulation in coronary artery disease (CAD) patients and healthy age-matched controls during rest and acute laboratory stress.

DETAILED DESCRIPTION:
BACKGROUND:

The strong association between mental stress and morbid cardiovascular events in coronary artery disease (CAD) patients may derive from stress-induced cardiac ischemia due to exaggerated increases in vascular resistance and arterial pressure. In fact, this may explain part of the prognostic relationship of baroreflex cardiac vagal control to cardiovascular outcome among CAD patients. The hemodynamic responses to psychological stress are buffered by the arterial baroreflex; thus, exaggerated pressor responses to mental stress may result from impaired baroreflex regulation in CAD patients.

DESIGN NARRATIVE:

The study has three components. The first component characterizes the relationships between vascular stiffness and baroreflex regulation among CAD patients, also contrasting healthy control subjects with CAD patients. The second component examines, in relation to individual differences in pharmacologically derived estimates of baroreflex function, changes in autonomic and baroreflex control during laboratory psychological stress among CAD patients and among healthy control subjects. The third component tests the hypothesis that impaired baroreflex regulation in CAD patients, due to increased vascular stiffness and/or attenuated autonomic control, is associated with exacerbated hemodynamic reactions to psychological stress. Bolus vasoactive drug infusions in combination with Finapres beat-by-beat arterial pressures and carotid B-mode ultrasonography are used to evaluate baroreflex sensitivity and arterial stiffness. Baroreflex adjustments to psychological stress are assessed by power spectral-derived relations between arterial pressure and cardiac chronotropy during a mental arithmetic task and a speech task. The degree to which indices of baroreflex function are associated with hemodynamic responses to psychological stress among CAD patients is assessed.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Taylor — Hebrew Rehabilitation Center for Aged

REFERENCES:
- [Background] Lipman RD, Grossman P, Bridges SE, Hamner JW, Taylor JA. Mental stress response, arterial stiffness, and baroreflex sensitivity in healthy aging. J Gerontol A Biol Sci Med Sci. 2002 Jul;57(7):B279-84. doi: 10.1093/gerona/57.7.b279. PMID 12084798
- [Background] Lipman RD, Salisbury JK, Taylor JA. Spontaneous indices are inconsistent with arterial baroreflex gain. Hypertension. 2003 Oct;42(4):481-7. doi: 10.1161/01.HYP.0000091370.83602.E6. Epub 2003 Sep 15. PMID 12975383
- [Background] Hunt BE, Farquhar WB. Nonlinearities and asymmetries of the human cardiovagal baroreflex. Am J Physiol Regul Integr Comp Physiol. 2005 May;288(5):R1339-46. doi: 10.1152/ajpregu.00038.2004. Epub 2005 Mar 3. PMID 15746307